CLINICAL TRIAL: NCT03942237
Title: Transmuscular Quadratus Lumborum Block for Postoperative Pain After Laparoscopic Adrenalectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Cui Xulei, Attending physician, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: cuixulei8
Record Dates: First submitted 2019-05-07; First posted 2019-05-08 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Pain Management; Nerve Block; Laparoscopic Adrenalectomy
Keywords: transmuscular quadratus lumborum block; adrenalectomy
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- single-injection QLB (quadratus lumborum block) (Experimental): Single-injection of QLB with local anesthetic is given preoperatively
  Interventions: Procedure: single-injection QLB(quadratus lumborum block)
- Placebo control (Placebo Comparator): Single-injection of QLB with NS is given preoperatively
  Interventions: Procedure: Placebo Control

INTERVENTIONS:
Procedure: single-injection QLB(quadratus lumborum block) — Inject 0.4ml/kg 0.5% ropivacaine between quadratus lumborum and psoas major muscle
  Device: The curved (C1-5) probe of Ultrasound Scanner Philips CX50 is used for scan
  Drug: single dose ropivacaine 0.4ml/kg 0.5% ropivacaine is given immediately after the correct position of needle tip is verified.
  Arms: single-injection QLB (quadratus lumborum block)
Procedure: Placebo Control — Inject 0.4ml/kg saline between quadratus lumborum and psoas major muscle
  Device: The curved (C1-5) probe of Ultrasound Scanner Philips CX50 is used for scan
  Drug: single dose 0.4ml/kg 0.9% NS is given immediately after the correct position of the needle tip is verified
  Arms: Placebo control

SUMMARY:
This prospective, randomized control study aims to compare the analgesic effect, satisfaction with anesthesia and analgesia between single-injection QLB (quadratus lumborum block)+general anesthesia (GA) and general anesthesia (GA) alone in patients undergoing laparoscopic adrenalectomy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 yrs
* American Society of Anesthesiologists physical statusⅠ-Ⅲ
* Undergo laparoscopic adrenalectomy
* Informed consent

Exclusion Criteria:

* a known allergy to the medications being used for anesthesia
* coagulopathy or on anticoagulants
* chronic opioid therapy or history of substance abuse
* participating in another RCT
* inability to properly describe postoperative pain to investigators (e.g., language barrier, neuropsychiatric disorder).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2019-08-28 (Actual); Study Completion 2019-09-02 (Actual)

PRIMARY OUTCOMES:
the NRS pain scores on activity 12-hours after surgery | 12-hours after surgery
  The NRS (a number scale from 0 to 10) is a commonly used pain intensity rating tool

SECONDARY OUTCOMES:
the pain scores at rest determined by the numeric rating scale (NRS, 0-10) | At 2,4, 8, 12, 24 ,48,72 hours after the surgery
  The NRS (a number scale from 0 to 10) is a commonly used pain intensity rating tool
incidence of postoperative nausea and vomiting (PONV) | within 24 postoperative hours
ambulation time | within 5 days after surgery
time of recovery of bowel movement | within 5 days after surgery
  defined as the time to first flatus
postoperative length of hospital stay | up to 2 weeks after surgery
patient's satisfaction of anesthesia and analgesia | 48 hours after surgery
  use the Chinese version of Bauer questionnaire to assess the patient satisfaction of anesthesia
the NRS pain scores on activity after surgery | At 2,4, 8, 24 ,48,72 hours after the surgery
  The NRS (a number scale from 0 to 10) is a commonly used pain intensity rating tool

CONTACTS AND LOCATIONS:
Overall Officials: Yuguang Huang, Study Chair — PUMCH
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

REFERENCES:
- [Derived] Yuan Q, Lu S, Cui X, Zhang Y, Xie Y, Zhang Y, Yan W, Ji Z, Huang Y. Transmuscular quadratus lumborum block for postoperative pain and recovery after laparoscopic adrenalectomy: a randomized controlled trial. BMC Anesthesiol. 2021 Nov 9;21(1):274. doi: 10.1186/s12871-021-01494-4. PMID 34753425